CLINICAL TRIAL: NCT06906328
Title: MEthylphenidate in ADHD - Addiction(s) Comorbidity: Value of Adding a Cognitive Remediation Program to Improve Short- and Medium-term Therapeutic Response
Acronym: META
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC23_0506
Record Dates: First submitted 2025-01-23; First posted 2025-04-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: ADHD-add
Keywords: Methylphenidate; Cognitive remediation; Functional improvement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive remediation program (Experimental): The cognitive remediation program under study (experimental treatment) consists of cognitive exercises performed on computers, in 30-45 minute sessions. The cognitive exercises target the deficits commonly observed in ADHD, a fortiori when it is associated with addictive disorders (working memory, inhibitory control, cognitive flexibility, attention, planning). The proposed program will be based on a software solution for cognitive rehabilitation, developed and validated for the treatment of attention and memory disorders and neurodegenerative, neurotraumatic and neuropsychiatric pathologies (PRESCO® software, marketed by HappyNeuron).
  Interventions: Behavioral: Cognitive remediation program, with the PRESCO® software
- Control program (Active Comparator): For the control program (comparator), we will use a software solution from the same company, but dedicated to stimulating and training auditory functions (AUDITICO® software). The advantage of this solution is that, like PRESCO®, it offers training exercises that are not aimed at re-educating cognitive functions. These include, for example, sound identification and discrimination activities. This tool can also be used by anyone, and is accessible for follow-up by the practitioner. It also offers levels of increasing difficulty, making it stimulating for users.
  Interventions: Behavioral: Control program, with the AUDITICO® software

INTERVENTIONS:
Behavioral: Cognitive remediation program, with the PRESCO® software — The program runs for 12 weeks, with two sessions per week, one with a neuropsychologist. In the first 4 weeks, the patient will have weekly sessions at the center and complete the other session at home using the app provided for the study. For the next 8 weeks, sessions with the neuropsychologist will be every other week, with the other session at home. The neuropsychologist will track progress through the software history and follow up by phone if needed.
  The proposed program will be based on a software solution for cognitive rehabilitation, developed and validated for the treatment of attention and memory disorders and neurodegenerative, neurotraumatic and neuropsychiatric pathologies (PRESCO® software, marketed by HappyNeuron).
  Arms: Cognitive remediation program
Behavioral: Control program, with the AUDITICO® software — Control program, with the same functional characteristics but without the targeted cognitive functions.
  For the control program (comparator), we will use a software solution from the same company, but dedicated to stimulating and training auditory functions (AUDITICO® software). The advantage of this solution is that, like PRESCO®, it offers training exercises that are not aimed at re-educating cognitive functions. These include, for example, sound identification and discrimination activities. This tool can also be used by anyone, and is accessible for follow-up by the practitioner. It also offers levels of increasing difficulty, making it stimulating for users.
  Arms: Control program

SUMMARY:
MEthylphenidate in ADHD - Addiction(s) comorbidity: benefit of adding a cognitive remediation program to improve short- and medium-term therapeutic response

DETAILED DESCRIPTION:
It seems essential to optimize the therapeutic management of patients suffering from ADHD/addiction(s) comorbidity by specifically targeting their neuropsychological deficits, in addition to the pharmacological and psychosocial approaches currently recommended. By intensively training deficient functions on the one hand, and promoting the development of compensatory strategies on the other, cognitive remediation could thus be a therapeutic tool of choice, producing beneficial effects that persist over time and translate into objectifiable changes in daily life. Cognitive training programs have been successfully proposed to patients with ADHD, but these were mainly programs designed for children, and very few studies have been carried out in adults, a fortiori in adults with ADHD-addiction(s) comorbidity.

The main aim of the study was to evaluate the effectiveness of cognitive remediation compared with the control program in addition to MPH treatment in reducing the functional impact of ADHD in patients with other addictive comorbidities, at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age over 15 (patients treated in the "adult" stream);
* Diagnosis of ADHD confirmed by DIVA-5 interview (for patients over 18) or Young DIVA-5 (for patients between 15 and 17) following a specialized ADHD-addiction(s) consultation;
* Indication for MPH treatment according to European recommendations (J. J. S. Kooij et al., 2019) and absence of contraindications (particularly cardiological);
* Presence of at least one comorbid addictive disorder (TUS and/or AC);
* Having given their consent to take part in the study;
* Being affiliated to the French social security system or benefiting from such a system.

Exclusion Criteria:

* Presence of disorders of the higher functions or difficulties in reading or writing the French language making it impossible to collect data;
* Pregnant or breast-feeding woman;
* Person deprived of liberty;
* Person under compulsory psychiatric care;
* Participation in another interventional research protocol involving another psychotherapeutic or pharmacological intervention that may have an impact on clinical outcome;
* Guardianship or safeguard of justice.

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2028-12-11 (Estimated); Study Completion 2029-12-11 (Estimated)

PRIMARY OUTCOMES:
Immediate ADHD functional improvement, at the end of the CRT (Cognitive remediation therapy) program | 9 month
  Evaluate the effectiveness of cognitive remediation versus the control program, alongside MPH treatment, in reducing the functional impact of ADHD in patients with addictive comorbidities at the end of treatment
  Functional improvement can be defined as an improvement of at least 30% in the functional impact score between post- and pre-treatment assessment. In our study, the functional outcome score used will be the global score of the WFIRS (Weiss Functional Impairment Rating Scale, A score of more than 1.5 points is considered to be representative of an impairment in the area concerned. Higher scores mean a worse outcome, the minimum and maximum values for each score are 0 and 3 respectively) questionnaire. The primary endpoint will therefore be the proportion of patients achieving functional improvement (at least 30% improvement in WFIRS score) in each group, estimated at the end of treatment.

SECONDARY OUTCOMES:
Sustained ADHD functional improvement, 6 months after the end of CRT. | 9 month
  To evaluate the efficacy of cognitive remediation compared with the control program in addition to MPH treatment in reducing the functional impact of ADHD in patients with other addictive comorbidities, 6 months after the end of treatment
  The endpoint will be the proportion of patients achieving functional improvement (at least 30% improvement in WFIRS score (Weiss Functional Impairment Rating Scale, A score of more than 1.5 points is considered to be representative of an impairment in the area concerned. Higher scores mean a worse outcome, the minimum and maximum values for each score are 0 and 3 respectively)) in each group, estimated 6 months after the end of treatment.
Immediate and sustained ADHD symptom improvement, both at the end of CRT and 6 months later. | 9 month
  To evaluate the efficacy of cognitive remediation versus the control program, alongside MPH treatment, in reducing ADHD symptoms in patients with comorbid addictions, at the end of treatment and 6 months post-treatment
  The evaluation criterion will be the proportion of patients who achieved symptom improvement (at least 30% improvement in the ASRS score (Adult ADHD Self-Report Scale Symptom Checklist, higher scores mean a worse outcome, the minimum and maximum values for each score are 0 and 36 respectively) for the dominant ADHD subtype, or either in case of combined type) in each group, estimated at treatment end or 6 months later.
Immediate and sustained improvement of neuropsychological deficits, both at the end of CRT and 6 months later. | 9 month
  To compare the efficacy of cognitive remediation versus the control program in addition to MPH treatment, at the end of treatment and 6 months after the end of treatment, in improving neuropsychological deficits.
  Neuropsychological deficits will be evaluated using performance scores on a series of neurocognitive tasks assessing key cognitive functions (all performance scores will be standardized to be comparable, i.e. Z-scores):
  * D2-R (selective attention),
  * Digit memory test (short-term memory and working memory),
  * Stroop test (inhibition),
  * Verbal fluency test (spontaneous flexibility)
  * Zoo test (planning)
Immediate and sustained improvement of the severity of comorbid addictive disorders, both at the end of CRT and 6 months later. | 9 month
  To compare the efficacy of cognitive remediation versus the control program in addition to MPH treatment, at the end of treatment and 6 months after the end of treatment, in reducing the severity of comorbid addictive disorders
  The severity of comorbid addictive disorders will be assessed based on the number of diagnostic criteria met in the diagnostic interviews, including:
  * MINI-S (alcohol and substance use disorders),
  * NODS (gambling disorder),
  * Diagnostic interview adapted from NODS for sexual addiction,
  * Diagnostic interview adapted from NODS for gaming disorder,
  * YFAS for food addiction,
  * Mc Elroy for compulsive buying.
Immediate and sustained improvement of the psychopathological characteristics associated with ADHD-addiction(s) comorbidity, both at the end of CRT and 6 months later. | 9 month
  Compare the efficacy of cognitive remediation versus the control program, in addition to MPH treatment, at the end of treatment and 6 months later, in alleviating psychopathological features associated with ADHD-addiction(s) comorbidity. Psychopathological characteristics associated with ADHD-addiction(s) comorbidity will be assessed by (all scores will be standardized to be comparable, i.e. Z-scores):
  * UPPS-P (Urgency, Premeditation (lack of), Perseverance (lack of), Sensation seeking impulsivity behavior scale, higher scores mean a worse outcome, the minimum and maximum values for each score are 4 and 16 respectively), (impulsivity): 5 scores,
  * DERS-16(Difficulties in Emotion Regulation Scale, higher scores mean a worse outcome, the minimum and maximum values are 16 and 80 respectively), (emotional dysregulation): 5 scores,
  * RSES (Rosenberg Self-Esteem Scale, higher score mean a better outcome, the minimum and maximum values are 10 and 40 respectively), (self-esteem): 1 score.
Immediate and sustained improvement of adherence to MPH treatment, both at the end of CRT and 6 months later. | 9 month
  To compare the efficacy of cognitive remediation versus the control program in addition to MPH treatment, at the end of treatment and 6 months after the end of treatment, in enhancing adherence to MPH treatment through CRT.
  Adherence to treatment will be evaluated based on:
  * Compliance with and tolerance to medication (structured interview, vital signs, and weight checks at follow-up visits)
  * The number of CRT sessions completed relative to the number of planned sessions.
Immediate and sustained ADHD functional improvement, both at the end of CRT and 6 months later, compared between ADHD subtypes (predominantly inattentive, predominantly impulsive/hyperactive, or combined type) | 9 month
  To analyze the short- and medium-term evolution of functional impairment based on ADHD subtype (predominantly inattentive, predominantly impulsive/hyperactive, or combined type).
  Functional impairment will be assessed using the WFIRS (Weiss Functional Impairment Rating Scale, A score of more than 1.5 points is considered to be representative of an impairment in the area concerned. Higher scores mean a worse outcome, the minimum and maximum values for each score are 0 and 3 respectively), (improvement of at least 30% in the functional impact score between post- and pre-treatment assessment), and the ADHD subtype will be determined using the DIVA-5 diagnostic interview.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHRU Brest, Brest, Brittany Region
  - EPSM du Finistère Sud, Quimper, Brittany Region
  - EPSM Georges Daumézon (Fleury-les-Aubrais, Loiret), Fleury-les-Aubrais, Centre-Val de Loire
  - CHRU de Tours, Tours, Centre-Val de Loire
  - CH Georges Daumézon - Bouguenais, Bouguenais, Loire-Atlantique
  - CHU Nantes, Nantes